CLINICAL TRIAL: NCT01433263
Title: A Randomized, Double-blind, Placebo-controlled Multi-center Study of BYM338 for Treatment of Cachexia in Patients With Stage IV Non-small Cell Lung Cancer or Stage III/IV Adenocarcinoma of the Pancreas
Brief Title: Clinical Study of BYM338 for the Treatment of Unintentional Weight Loss in Patients With Cancer of the Lung or the Pancreas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CBYM338X2202
Record Dates: First submitted 2011-08-24; First posted 2011-09-13 (Estimated); Results first posted 2015-05-13 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2016-02

CONDITIONS: Cachexia
Keywords: Wasting syndrome; emaciation; lung cancer; adenocarcinoma; pancreatic cancer
MeSH Terms: conditions — Cachexia; Wasting Syndrome; Emaciation; Lung Neoplasms; Adenocarcinoma; Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 30mg/kg BYM338 (Experimental)
  Interventions: Drug: BYM338 active drug
- Placebo / late 30mg/kg BYM338 (Placebo Comparator)
  Interventions: Drug: BYM338 active drug; Drug: Placebo

INTERVENTIONS:
Drug: BYM338 active drug
Drug: Placebo
  Arms: Placebo / late 30mg/kg BYM338

SUMMARY:
A safety & efficacy clinical study of the investigational medicinal product BYM338 for the treatment of unintentional weight loss in patients with cancer of the lung or the pancreas

ELIGIBILITY:
Key Inclusion criteria:

1. Patients must sign an informed consent before assessment
2. Patients with pathologically and/or clinically confirmed diagnosis of stage IV non-small (squamous or non-squamous) cell lung cancer (NSCLC) or stage III/IV adenocarcinoma of the pancreas.
3. Patients with stage IV NSCLC will be receiving or completed or discontinued standard chemotherapy or be chemotherapy-naive by choice.
4. Patients with stage III/IV pancreatic adenocarcinoma will be receiving standard chemotherapy or no chemotherapy. If patients are receiving chemotherapy, a change in chemotherapy is not expected.
5. Greater than or equal to 5% unintentional weight loss over the previous 3-6 months, not explained by simple starvation. Simple starvation is considered to be excluded when weight loss is not ameliorated by standard nutritional counseling and oral supplementation over a 2 week period.
6. Body mass index (BMI) ≤ 30 kg/m2.
7. Life expectancy of at least 4 months.
8. Able to communicate well and comply with the requirements of the study, including by phone and written logs.

Key Exclusion criteria:

1. Patients who have received investigational anti-neoplastic therapy within 3 weeks of screening
2. Evidence of inadequate organ or brain function, as defined by lab tests and imaging
3. Patients with severe and/or uncontrolled medical conditions that could interfere with the study (e.g. heart conditions, high blood pressure, diabetes, infection) uncontrolled pain or any other non-stable illness
4. Pregnant or lactating women.
5. Women capable of becoming pregnant must use highly effective contraception during the study and for 8 weeks after stopping treatment. All female patients must have negative pregnancy test results throughout the study
6. Patients unwilling or unable to follow instructions.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2011-08; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- United States (6):
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, San Antonio, Texas
- Novartis Investigative Site, Vilnius, Lithuania
- Novartis Investigative Site, Bucharest, Romania
- Novartis Investigative Site, Sankt Gallen, Switzerland
- Novartis Investigative Site, Edinburgh, United Kingdom

REFERENCES:
- [Derived] Epstein SA, Doles JD, Dasgupta A. KLF10: a point of convergence in cancer cachexia. Curr Opin Support Palliat Care. 2024 Sep 1;18(3):120-125. doi: 10.1097/SPC.0000000000000711. Epub 2024 Jul 15. PMID 39007915

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Core Phase single dose BYM338 30mg/kg i.v. active or placebo with 8week followup. Followup phase started Week 8 & patients on placebo in the Core Phase were given BYM338 & patients on BYM338 in Core Phase continued to be followed for an additional 8 weeks. Late BYM338 are patients who received Placebo during Core Phase and then BYM338 after Week 8.
Period: Overall Study
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Started | 29 | 28
Completed | 10 | 16
Not Completed | 19 | 12
Not completed — Adverse Event | 3 | 1
Not completed — Death | 5 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Deviation | 1 | 0
Not completed — Withdrawal by Subject | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338 | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.17) | 61.5 (10.74) | 62.1 (10.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline of Thigh Muscle Volume (TMV) by MRI Scan at Week 8
Description: Thigh Muscle Volume (TMV) change was evaluated by a responder analysis. Patients whose loss of muscle TMV by MRI was no more than or equal to 2% at Week 8 was considered responders.
Time Frame: Baseline, week 8
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data. However, for a given time frame, analyzed participants had values at both baseline and the corresponding time frame, i.e. week 8
Measure: Mean (Standard Deviation); unit: Percentage Change of TMV
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 15 | 22
Percentage Change of TMV | 2.0 (8.094) | 0.65 (8.239)

2. Secondary Outcome: Percentage Change in Body Weight From Baseline at Week 7 and Week 9
Description: Percentage Change in body weight from baseline in killograms (kg) at week 7 and week 9
Time Frame: Baseline, Week 7 and Week 9
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data.
Measure: Mean (Standard Deviation); unit: Percent Change of Weight (kg)
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 29 | 28
Percent Change of Weight (kg)
  Week 7 (n= 15, 17) | -3.3 (5.035) | -0.68 (4.457)
  Week 9 (n=14,16) | -1.8 (7.131) | -0.32 (3.271)

3. Secondary Outcome: Maximum Observed Serum Concentration (Cmax)
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn on Day 1 30mg/kg BYM338 (Core)or week 8 Late 30mg/kg BYM338 (when placebo subjects were rolled over to active). PK parameters were calculated from plasma concentration-time data using non-compartmental methods.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Day 1 and Week 8
Population: Pharmacokinetics (PK) analysis set: Patients with evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 29 | 14
ng/ml | 422 (142) | 408 (78.4)

4. Secondary Outcome: Time to Reach the Maximum Concentration After Drug Administration (Tmax)
Description: Blood samples for pharmacokinetic (PK) evaluation were drawn on Day 1 30mg/kg BYM338 (Core)or week 8 Late 30mg/kg BYM338 (when placebo subjects were rolled over to active). Tmax was directly determined from the raw serum concentration-time data.
Time Frame: 0, 1, 2, 3, 4, 6, 8, 12, 24, 48, 72, 96 hours post-dose on Day 1 and Week 8
Population: Pharmacokinetics (PK) analysis set: Patients with evaluable PK data.
Measure: Median (Inter-Quartile Range); unit: hr
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 29 | 14
hr | 2.05 (142) [1.83 to 3.92] | 2.22 (78.4) [2.00 to 4.00]

5. Secondary Outcome: Percentage Change From Baseline in Total Lean Body Mass (LBM) by Dual-Energy X-ray Absorptiometery (DXA) Compared to Placebo: at Week 8
Description: total lean body mass (LBM) is measured by dual energy x-ray absorptiometry (DXA).Percent Change = [(LBM at Visit - LBM at Baseline) / LBM at Baseline] * 100.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage Change in LBM
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 19 | 22
Percentage Change in LBM | 4.97 (7.537) | 2.41 (4.625)

6. Secondary Outcome: Percentage Change From Baseline of Bone Mineral Density (BMD) by Dual-Energy X-ray Absorptiometery (DXA) Compared to Placebo at Week 8
Description: Bone Mineral Density (BMD)is measured by dual energy x-ray absorptiometry (DXA).Percent Change = [(BMD at Visit - BMD at Baseline) / BMD at Baseline] * 100.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage Change in BMD
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 19 | 22
Percentage Change in BMD | 0.51 (3.712) | 0.14 (4.14)

7. Secondary Outcome: Percentage Change From Baseline of Physical Activity Levels (Using the ActivPAL™ Device) Number of Steps Taken Compared to Placebo at Week 4 and 7
Description: Each patient was required to wear the ActivPal™ for a span of 6 days at Week 4 and Week 7 for patient home activity recording. The ActivPal™ was given to patients in clinic to wear for 6 consecutive days. The ActivPAL™ records periods spent sitting, standing and walking, sit-to-stand transitions, step count and rate of stepping (cadence) over a maximum period of 10 days with a fully charged new battery.
Time Frame: Baseline, Week 4 and Week 7
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data.
Measure: Mean (Standard Deviation); unit: percentage change in number of steps
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 27 | 28
percentage change in number of steps
  Week 4 (n=18, 23) | 917.78 (3720.491) | 63.59 (130.913)
  Week 7 (n=13, 22) | -17.37 (80.350) | 35.80 (119.486)

8. Secondary Outcome: Percentage Change From Baseline of Physical Activity Levels (Using the ActivPAL™ Device) Time Sedentary Taken Compared to Placebo at Week 4 and 7
Description: as for outcome 7
Time Frame: Baseline, Week 4 and Week 7
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data.
Measure: Mean (Standard Deviation); unit: percentage change in time (minutes)
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 27 | 28
percentage change in time (minutes)
  Week 4 (n=18, 23) | -0.05 (10.049) | 52.25 (207.403)
  Week 7 (n=13, 22) | 107.85 (280.791) | 60.25 (222.366)

9. Secondary Outcome: Percentage Change From Baseline of Physical Activity Levels (Using the ActivPAL™ Device) Time Standing Compared to Placebo at Week 4 and 7
Description: as for outcome 7
Time Frame: Baseline, Week 4 and Week 7
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data.
Measure: Mean (Standard Deviation); unit: percentage change in time (minutes)
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 27 | 28
percentage change in time (minutes)
  Week 4 (n=18, 23) | 1.82 (78.364) | 38.17 (111.361)
  Week 7 (n=13, 22) | 41.90 (251.291) | 23.76 (99.268)

10. Secondary Outcome: Percentage Change From Baseline of Physical Activity Levels (Using the ActivPAL™ Device) Time Stepping Compared to Placebo at Week 4 and 7
Description: as for outcome 7
Time Frame: Baseline, Week 4 and Week 7
Population: Pharmacodynamics (PD) analysis set: Patients with evaluable PD parameter data.
Measure: Mean (Standard Deviation); unit: percentage change in time (minutes)
Arm/Group | 30mg/kg BYM338 | Placebo / Late 30mg/kg BYM338
Number analyzed (Participants) | 27 | 28
percentage change in time (minutes)
  Week 4 (n=18, 22) | 1446.69 (6011.324) | 85.30 (159.949)
  Week 7 (n=13, 21) | -31.64 (67.180) | 33.39 (129.218)

ADVERSE EVENTS:
Groups:
- Core - 30mg/kg BYM338: Core - 30mg/kg BYM338
- Core - Placebo: Core - Placebo
- Follow-up - 30mg/kg BYM338: Follow-up - 30mg/kg BYM338
- Follow-up - Placebo: Follow-up - Placebo
- Follow-up - 30mg/kg BYM338 Late: Follow-up - 30mg/kg BYM338 Late
Arm/Group | Core - 30mg/kg BYM338 | Core - Placebo | Follow-up - 30mg/kg BYM338 | Follow-up - Placebo | Follow-up - 30mg/kg BYM338 Late
Serious Adverse Events (participants affected / at risk) | 18/29 | 4/28 | 7/19 | 1/3 | 7/21
Other Adverse Events (participants affected / at risk) | 19/29 | 19/28 | 12/19 | 2/3 | 13/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Core - 30mg/kg BYM338 (N=29) | Core - Placebo (N=28) | Follow-up - 30mg/kg BYM338 (N=19) | Follow-up - Placebo (N=3) | Follow-up - 30mg/kg BYM338 Late (N=21)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Klebsiella infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 0 | 3 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Angiopathy (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Core - 30mg/kg BYM338 (N=29) | Core - Placebo (N=28) | Follow-up - 30mg/kg BYM338 (N=19) | Follow-up - Placebo (N=3) | Follow-up - 30mg/kg BYM338 Late (N=21)
Anaemia (Blood and lymphatic system disorders) | 4 | 6 | 2 | 1 | 3
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 2 | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 2 | 1 | 1 | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 3 | 1 | 0 | 5
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 5 | 1 | 0 | 0 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 2
Asthenia (General disorders) | 2 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 6 | 3 | 4 | 1 | 1
Oedema peripheral (General disorders) | 3 | 3 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 2 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0
Candida infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0
Gingival infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 2
Blood bilirubin increased (Investigations) | 1 | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 1 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 1 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 4 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 1 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Benign neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 2
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 1 | 0 | 0 | 2
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0 | 0
Bladder irritation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial